CLINICAL TRIAL: NCT00167479
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Risperidone Monotherapy in Ambulatory Bipolar Disorder With Current at Least Moderately Severe Anxiety and Lifetime Panic Disorder or Generalized Anxiety Disorder
Brief Title: A Study of Risperidone Monotherapy in Bipolar Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101541d; RIS-BIP-408
Record Dates: First submitted 2005-09-10; First posted 2005-09-14 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Bipolar Disorder; Panic Disorder; Generalized Anxiety Disorder
Keywords: Bipolar Anxiety; Bipolar Disorder; Anxiety; Panic Disorder; Generalized Anxiety Disorder; GAD; Risperidone; Double-Blind; Placebo Controlled
MeSH Terms: conditions — Bipolar Disorder; Panic Disorder; Generalized Anxiety Disorder; Anxiety Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone (Risperdal)

SUMMARY:
The specific aim of this study is to evaluate the efficacy, tolerability, and safety of risperidone monotherapy in the treatment of ambulatory bipolar disorder with comorbid lifetime panic disorder or generalized anxiety disorder and current at least moderately severe anxiety.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, parallel-group, 8-week trial of risperidone monotherapy in outpatient subjects with a lifetime bipolar I, II, or NOS disorder, a lifetime panic or generalized anxiety disorder, and current at least moderately severe anxiety symptoms. Approximately 90 subjects will be enrolled to obtain 60 subjects who complete the 8-week trial. Subjects will be randomized to risperidone or placebo in a 1:1 ratio. No concomitant psychotropic medication will be allowed except for prn lorazepam during the first two weeks for the management of affective and anxiety symptoms, and prn zolpidem and zaleplon throughout the study for the management of insomnia. Throughout the study, psychiatric scales will be used to assess psychiatric symptoms and the presence of treatment-emergent adverse events will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older.
2. Subjects must have lifetime bipolar I, II, or NOS disorder as defined by DSM-IV criteria.
3. Subjects must have lifetime panic disorder or generalized anxiety disorder (GAD) as defined by DSM-IV criteria (except clause "does not occur exclusively during a mood disorder" of Criterion F for GAD) .
4. Subjects' bipolar symptoms must be no more than moderately severe, defined as a CGI-BP < 4.
5. Subjects' anxiety symptoms must be at least moderately severe, defined as a CGI-S > 4.
6. Subjects must not be receiving mood stabilizing, antidepressant, antipsychotic, or anxiolytic medication for > one week prior to baseline. Patients receiving fluoxetine or depot antipsychotics should be off these medications for > four weeks prior to baseline.
7. Subjects or their legally authorized representative must sign the Informed Consent Document after the nature of the trial has been fully explained.
8. If female, subjects must be: postmenopausal, surgically incapable of childbearing, or practicing medically acceptable effective method(s) of contraception (e.g., hormonal methods, double barrier methods, intrauterine device) for at least one month prior to study entry and throughout the study.

Exclusion Criteria:

1. Subjects who do not have lifetime bipolar disorder by DSM-IV-TR criteria.
2. Subjects who do not have lifetime panic disorder or generalized anxiety disorder by DSM-IV-TR criteria.
3. Subjects who are receiving treatment with an antimanic or mood stabilizing medication (lithium, valproate, carbamazepine, or an antipsychotic), and in the investigators' judgment, require ongoing treatment with that medication.
4. Subjects whose bipolar symptoms are presently more than moderately severe (CGI-BP > 5).
5. Subjects whose anxiety symptoms are presently less than moderately severe (CGI < 3).
6. Subjects with clinically significant suicidal or homicidal ideation.
7. Subjects with current psychotic symptoms.
8. Subjects with a current DSM-IV Axis I diagnosis of delirium, dementia, amnesia, or other cognitive disorders; a DSM-IV diagnosis of a substance dependence disorder within the past six months; a lifetime DSM-IV psychotic disorder (e.g., schizophrenia or schizoaffective disorder).
9. Subjects with serious general medical illnesses including hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, or hematologic disease as determined by the clinical judgment of the clinical investigator. Subjects with hypo- or hyperthyroidism unless stabilized on thyroid replacement > 3 months.
10. Subjects with a clinically significant abnormality in their prestudy physical exam, vital signs, EKG, or laboratory tests.
11. Subjects who are allergic to or who have demonstrated hypersensitivity to risperidone.
12. Women who are pregnant or nursing.
13. Subjects who have received an experimental drug or used an experimental device within 30 days.
14. Subjects who have a history of neuroleptic malignant syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-09; Study Completion 2006-09

PRIMARY OUTCOMES:
Clinician Global Improvement Scale (CGI-21)

SECONDARY OUTCOMES:
Sheehan Panic Disorder Scale (SPS)
The Psychic and Somatic factors of the HAM-A
Young Mania Rating Scale, Total Score
Inventory of Depressive Symptoms, Total Score
Patient Global Improvement Scale (PGI-21)
The Clinician Global Improvement-Bipolar (CGI-BP)
The Family Impact Scale (FIS)
The Sheehan Disability Scale - Total Disability Score, Work Disability Score, Social Disability Score, Family Disability Score

CONTACTS AND LOCATIONS:
Overall Officials: David V. Sheehan, MD, MBA, Principal Investigator — University of South Florida College of Medicine; Susan L. McElroy, MD, Principal Investigator — University of Cincinatti, Department of Psychiatry; Trisha - Suppes, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center; Paul E. Keck, MD, Principal Investigator — University of Cincinatti, Department of Psychiatry
Locations (3):
- United States (3):
  - University of South Florida Psychiatry Center, Tampa, Florida
  - University of Cincinatti, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas